CLINICAL TRIAL: NCT01169480
Title: The Impact of Giving a Massage on Perceived Depression, Anxiety and Stress of Massage Therapists: A Randomized Clinical Trial
Brief Title: The Impact of Giving a Massage
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anne M. Jensen, Senior Researcher, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Massage Study - I
Record Dates: First submitted 2010-04-26; First posted 2010-07-26 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Mental State, Reported as Depression, Anxiety or Stress
Keywords: Massage; Therapist, Massage; DASS; Depression; Anxiety, State; Anxiety, Trait; Stress; Touch; Therapeutic Relationship
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage Giver (Experimental): Participants in the experimental group will be asked to give one 50-minute Swedish massage to another volunteer.
  Interventions: Behavioral: Give a massage
- Passive Controls (No Intervention): Participants in this arm will wait in a classroom (as usual) and do nothing out of their ordinary routines.

INTERVENTIONS:
Behavioral: Give a massage — Participants in this arm will give a 50-minute Swedish massage to a volunteer.
  Arms: Massage Giver

SUMMARY:
The aim of this study is to investigate if giving a massage impacts the mental state of a massage therapist, including depression, anxiety, and stress . It is speculated that feelings of depression, anxiety and stress will reduce following the giving of a massage.

DETAILED DESCRIPTION:
Background It is well established that massage is beneficial for musculoskeletal conditions such as low back pain1-3 and neck pain. In addition, massage has been shown to alleviate depressive symptoms and reduce state anxiety and perceived stress. Furthermore, the therapeutic benefits of touch itself are recognized for many conditions and in many stages of life.

Thus far all massage research has investigated the impact of massage on the massage client, or the receiver of the massage. No peer-reviewed study was found that reported any biopsychosocial effects on the giver of the massage, the massage therapist.

With touch therapies such as massage, it is impossible to touch without being touched oneself. Therefore, it is speculated that the giver of a touch therapy will also receive a therapeutic benefit. In fact, it has been reported anecdotally that massage therapists often feel "better" after they give a massage than before. Feelings of exhilaration, enhanced well-being, and improved energy are common.

The aim of this study is to investigate if giving a massage impacts the state of mind of massage therapists, including depression, anxiety, and stress.

Methods

Participants For this study, 22 participants who are massage therapists, students of massage or recent graduates will be recruited from the Parker School of Massage Therapy(PSMT). Participants will be included if they are healthy and aged between 18 and 65 years old, and excluded if they currently have any of the following conditions: contusion, fracture, inflammatory arthritides, peripheral neuropathy, or pregnancy. Of the eligible volunteers, ten participants will be randomly selected to the experimental group, while the other ten participants will act as controls. All interventions will occur in the PSMT.

Interventions Participants in the experimental group will be asked to give one 50-minute Swedish massage to another volunteer. Control participants will be asked to wait in a classroom (i.e. do nothing) for the same amount of time.

Objectives The aim of this study is to investigate if giving a massage impacts the mental state of a massage therapist, including depression, anxiety, and stress. It is speculated that feelings of depression, anxiety and stress will reduce following the giving of a massage.

Outcomes The primary assessment measure will be the Depression, Anxiety, Stress Scales (DASS). The DASS is a set of three self-report scales measuring the affective states of depression ("D"), anxiety ("A") and stress ("S"). Each of the 21 items is scored from "0" (Did not apply to me at all) to "3" (Applied to me very much or most of the time). A template is used to score the test and subscore is achieved for each of the three subcategories. Subscores can range from 0 to 28+, with normals being at the lower end of the range. The DASS was found to have adequate convergent and discriminant validity and good reliability, including test-retest reliability.

Secondary outcome measure will be the State-Trait Anxiety Inventory-II (STAI). The STAI is a self-report measure that assesses both state anxiety (i.e. feelings at present moment) and trait anxiety (i.e. general feelings). The 40 items are measured on a 4-point Likert scale (1=Almost Never to 4=Almost Always). Scores are obtained for each subscale (State and Trait Anxiety) with the higher scores indicating higher anxiety. The STAI has been shown to be valuable in both research and clinical settings, and has been found to have high internal consistency, and excellent test-retest reliability.

Sample Size Sample size estimation was performed based on the primary outcome measure, the DASS. A minimum change in the total DASS score of 10 points is predicted using results from a similar effectiveness studies. Using the DSS Research Sample Size Calculator Software http://www.dssresearch.com/toolkit/sscalc/size_a2.asp), and a 5% level of confidence a total of 22 participants (11 per group) would be required for a statistical power of 0.81. We do not anticipate any loss-to-follow up and thus have not made any further adjustment for attrition.

Randomization & Blinding Participants meeting the eligibility criteria will be pooled and a random drawing will determine which individuals will be in the experimental group and give the massage and which will act as controls. An independent assistant will perform the randomization process. Another independent assistant who is blind to group allocation will administer the assessment measures. Participants will be blind to group allocation for the duration of the study. While it is very difficult to blind participants when hands-on therapies are investigated, in this study this will be accomplished because giving a massage is a routine part of the day for these participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are currently massage therapists, massage student or recent massage school graduates,
* Aged 18 to 65 years,
* Fluent in English

Exclusion Criteria:

* Current bruising,
* Fracture,
* Inflammatory arthritides,
* Peripheral neuropathy,
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Perceived, self-reported stress, anxiety and depression | Immediately before the 50-minute masage
  The primary assessment measure will be perceived, self-reported stress, anxiety and depression as measured by the Depression, Anxiety, Stress Scales (DASS). The DASS is a set of three scales measuring the states of depression, anxiety and stress. Each of the 21 items is scored from "0" (Did not apply to me at all) to "3" (Applied to me very much or most of the time). A subscore is achieved for each of the three subcategories. Subscores can range from 0 to 28+. The DASS was found to have adequate convergent and discriminant validity and good reliability, including test-retest reliability.

SECONDARY OUTCOMES:
Perceived, self-reported state and trait anxiety | Immediately before the 50-minute massage
  Secondary outcome measure will be perceived, self-reported state and trait anxiety as measured by the State-Trait Anxiety Inventory-II (STAI). The STAI is a self-report measure that assesses both state anxiety and trait anxiety. The 40 items are measured on a 4-point Likert scale (1=Almost Never to 4=Almost Always). Scores are obtained for each subscale with the higher scores indicating higher anxiety. The STAI has been shown to be valuable in both research and clinical settings, and has been found to have high internal consistency,19 and excellent test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: M Jensen, DC, MS, MSc, Study Director — Parker Research Institute; Lavada A Smith, PhD, Principal Investigator — Parker College School of Massage; Drew Riffe, DC, Study Chair — Parker College School of Massage
Locations (1):
- Parker College School of Massage, Dallas, Texas, United States